CLINICAL TRIAL: NCT03932565
Title: Clinical Trial Study of Interventional Therapy Sequential With the Fourth-generation CAR-T Cells (IL7 and CCL19 or / and IL12) Targeting Nectin4/FAP in the Treatment of Advanced Malignant Solid Tumors With Nectin4-positive
Brief Title: Interventional Therapy Sequential With the Fourth-generation CAR-T Targeting Nectin4/FAP for Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Sixth Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Zhejiang Qixin Biotech (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lishui People's Hospital
Record Dates: First submitted 2019-04-27; First posted 2019-04-30 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Nectin4-positive Advanced Malignant Solid Tumor
MeSH Terms: interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The fourth-generation CAR-T therapy (Experimental): Clinical trial study of Interventional therapy sequential with the fourth-generation CAR-T cells (IL7 and CCL19 or / and IL12) targeting Nectin4/FAP in the treatment of advanced malignant solid tumors with Nectin4-positive .
  Interventions: Biological: CAR-T therapy for nectin4-positive malignant solid tumor

INTERVENTIONS:
Biological: CAR-T therapy for nectin4-positive malignant solid tumor — The Intravenous minimally invasive surgery combined with intratumoral injection of Nectin4/FAP-targeted the fourth-generation CAR-T cells (expressing IL7 and CCL19, or IL12) are used to treat Nectin4-positive advanced malignant solid tumors, maximally eliminating residual cancer cells and preventing recurrence.

SUMMARY:
According to the high expression of tumor cell-associated antigen Nectin4 in patients with solid tumors such as non-small cell lung cancer, breast cancer, ovarian cancer, bladder cancer, and pancreatic cancer, and in order to target FAP-positive CAFs in the tumor-associated stroma, the Intravenous minimally invasive surgery combined with intratumoral injection of Nectin4/FAP-targeted fourth-generation CAR-T cells (expressing IL7 and CCL19, or IL12) are used to treat Nectin4-positive advanced malignant solid tumors, maximally eliminating residual cancer cells and preventing recurrence.

DETAILED DESCRIPTION:
Currently, malignant tumors are the leading cause of death. Surgery, chemotherapy, radiation therapy, and targeted therapy have become the four foundations of cancer treatment for many years. With the development of science and technology, immunotherapy has become the "fifth pillar" of cancer treatment. The most hot topic in immunotherapy is CAR-T therapy. The basic principle of CAR-T therapy (chimeric antigen receptor-T cells) is mainly to use the patient's own immune cells to clear cancer cells. CAR is a core component of CAR-T, conferring T cell a HLA-independent way to recognize tumor antigens, allowing CAR-modified T cells to recognize a broader target than the natural T cell surface receptor TCR. The basic design of CAR includes a tumor associated antigen (TAA) binding region, an extracellular hinge region, a transmembrane region and an intracellular signaling region. The selection of target antigens is a key determinant of the specificity and effectiveness of CAR and the safety of genetically modified T cells themselves.

Nectin-4 is a type I transmembrane protein whose extracellular domain is composed of three Ig-like domains (V-C-C type), which together with cadherin participate in the formation and maintenance of adhesion junctions. Nectin-4 is ubiquitously expressed in human embryonic cells but is hardly expressed in normal adult tissues. Nectin-4 is highly expressed on the surface of breast cancer, bladder cancer, non-small cell lung cancer, and pancreatic cancer cells, and plays a key role in the occurrence, invasion and metastasis of these epithelial malignancies. In conclusion, Nectin-4 is one of the important targets for the diagnosis and treatment of many solid tumors. The antibody-conjugated drug Enfortumab Vedotin targeting Nectin-4 was highly effective in Phase I clinical trials in 81 advanced bladder cancers, and was awarded FDA breakthrough therapy in March 2018. Fibroblast activation protein (FAP) belongs to the serine protease family and is highly expressed on the surface of cancer-associat

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the requirements voluntarily participate in the study and sign the Informed Consent Form.
2. Age is 18 to 75 years old, gender is not limited; the Eastern Cancer Cooperative Group (ECOG) scores 0 to 3
3. Pathological diagnosis of malignant solid tumors.
4. Advanced malignant solid tumors meet the CSCO malignant tumor diagnosis and treatment guidelines (2018 version). (Flow or pathology shows that tumor cells express Nectin4 antigen and tumor-associated fibroblasts express FAP antigen)
5. Head magnetic resonance or CT examination showed no central invasion of malignant tumors.
6. Collection of peripheral blood mononuclear cells must be more than 2 weeks from radiotherapy and chemotherapy.
7. Peripheral blood neutrophils number ≥ 1000 / μl, platelets ≥ 50,000 / μl.
8. Heart, liver and kidney function: creatinine <2.5mg/dl; ALT (alanine aminotransferase) / AST (aspartate aminotransferase) <3 times lower than the upper limit of normal; total bilirubin <2.0mg/dl.
9. Cardiac ejection fraction (EF) ≥ 50%, echocardiography without pericardial effusion.
10. Have fertility must be willing to use contraceptive methods.
11. The expected survival period is more than 12 weeks.
12. No other malignant tumors, severe autoimmune diseases or congenital immunodeficiency, serious progressive infection, cranial nerve disorder or mental illness.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with uncontrollable active infections.
3. Patients with systemic steroids; recent or current use of inhaled steroids is not excluded.
4. Previously involved CAR-T cell therapies produced any uncontrolled disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-13 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events that are related to treatment | 2 years
  Safety and tolerability measured by occurrence of study related adverse effects defined by NCI-CTCAE v4.03

SECONDARY OUTCOMES:
2 year overall survival(OS) | 2 years
  To estimate 2 year overall survival(OS) after the fourth-generation CAR-T cells (IL7 and CCL19 or / and IL12) targeting Nectin4/FAP in the treatment of advanced malignant solid tumors with Nectin4-positive
3 year progression free survival (PFS) | 3 years
  To estimate 3 year progression free survival after the fourth-generation CAR-T cells (IL7 and CCL19 or / and IL12) targeting Nectin4/FAP in the treatment of advanced malignant solid tumors with Nectin4-positive

CONTACTS AND LOCATIONS:
Overall Officials: Bingmu Fang, M.D, Principal Investigator — Lishui Country People's Hospital
Locations (2):
- China (2):
  - The Sixth Affiliated Hospital of Wenzhou Medical University, Lishui, Zhejiang
  - Zhejiang QiXin Biotech, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang LC, Lo A, Scholler J, Sun J, Majumdar RS, Kapoor V, Antzis M, Cotner CE, Johnson LA, Durham AC, Solomides CC, June CH, Pure E, Albelda SM. Targeting fibroblast activation protein in tumor stroma with chimeric antigen receptor T cells can inhibit tumor growth and augment host immunity without severe toxicity. Cancer Immunol Res. 2014 Feb;2(2):154-66. doi: 10.1158/2326-6066.CIR-13-0027. Epub 2013 Nov 12. PMID 24778279
- [Background] Lo A, Wang LS, Scholler J, Monslow J, Avery D, Newick K, O'Brien S, Evans RA, Bajor DJ, Clendenin C, Durham AC, Buza EL, Vonderheide RH, June CH, Albelda SM, Pure E. Tumor-Promoting Desmoplasia Is Disrupted by Depleting FAP-Expressing Stromal Cells. Cancer Res. 2015 Jul 15;75(14):2800-2810. doi: 10.1158/0008-5472.CAN-14-3041. Epub 2015 May 15. PMID 25979873
- [Background] Joyce JA, Fearon DT. T cell exclusion, immune privilege, and the tumor microenvironment. Science. 2015 Apr 3;348(6230):74-80. doi: 10.1126/science.aaa6204. PMID 25838376
- [Background] Challita-Eid PM, Satpayev D, Yang P, An Z, Morrison K, Shostak Y, Raitano A, Nadell R, Liu W, Lortie DR, Capo L, Verlinsky A, Leavitt M, Malik F, Avina H, Guevara CI, Dinh N, Karki S, Anand BS, Pereira DS, Joseph IB, Donate F, Morrison K, Stover DR. Enfortumab Vedotin Antibody-Drug Conjugate Targeting Nectin-4 Is a Highly Potent Therapeutic Agent in Multiple Preclinical Cancer Models. Cancer Res. 2016 May 15;76(10):3003-13. doi: 10.1158/0008-5472.CAN-15-1313. Epub 2016 Mar 24. PMID 27013195
- [Background] Kraman M, Bambrough PJ, Arnold JN, Roberts EW, Magiera L, Jones JO, Gopinathan A, Tuveson DA, Fearon DT. Suppression of antitumor immunity by stromal cells expressing fibroblast activation protein-alpha. Science. 2010 Nov 5;330(6005):827-30. doi: 10.1126/science.1195300. PMID 21051638
- [Background] Lopez M, Ghidouche A, Rochas C, Godelaine D, Carrasco J, Colau D, Hames G, Montero-Julian FA, Coulie PG, Olive D. Identification of a naturally processed HLA-A*02:01-restricted CTL epitope from the human tumor-associated antigen Nectin-4. Cancer Immunol Immunother. 2016 Oct;65(10):1177-88. doi: 10.1007/s00262-016-1877-7. Epub 2016 Aug 11. PMID 27514672
- [Background] Targeting Nectin-4 in Bladder Cancer. Cancer Discov. 2017 Aug;7(8):OF3. doi: 10.1158/2159-8290.CD-NB2017-095. Epub 2017 Jun 20. PMID 28634245
- [Background] Tsiatas M, Grivas P. Immunobiology and immunotherapy in genitourinary malignancies. Ann Transl Med. 2016 Jul;4(14):270. doi: 10.21037/atm.2016.06.29. PMID 27563657
- [Background] Srivastava S, Riddell SR. Chimeric Antigen Receptor T Cell Therapy: Challenges to Bench-to-Bedside Efficacy. J Immunol. 2018 Jan 15;200(2):459-468. doi: 10.4049/jimmunol.1701155. PMID 29311388
- [Background] Mirzaei HR, Rodriguez A, Shepphird J, Brown CE, Badie B. Chimeric Antigen Receptors T Cell Therapy in Solid Tumor: Challenges and Clinical Applications. Front Immunol. 2017 Dec 22;8:1850. doi: 10.3389/fimmu.2017.01850. eCollection 2017. PMID 29312333
- [Background] Adachi K, Kano Y, Nagai T, Okuyama N, Sakoda Y, Tamada K. IL-7 and CCL19 expression in CAR-T cells improves immune cell infiltration and CAR-T cell survival in the tumor. Nat Biotechnol. 2018 Apr;36(4):346-351. doi: 10.1038/nbt.4086. Epub 2018 Mar 5. PMID 29505028